CLINICAL TRIAL: NCT04567108
Title: SUBstituting With Preferred Options: Health Effects of Substituting Sugar-sweetened Beverages With Non-caloric Beverages in Adults With Overweight and Obesity
Brief Title: Health Effects of Substituting Sugary Beverages With Artificially-sweetened Beverages or Water
Acronym: SUB-POP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Deirdre K Tobias, ScD, Assistant Professor, Associate Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020p002494; 1R01DK125803-01 (NIH)
Record Dates: First submitted 2020-09-14; First posted 2020-09-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Body Weight
Keywords: Prevention; Weight control; Sugar-sweetened beverages; Artificial sweeteners; Water; Beverages
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Intervention Model Description: Parallel randomization on a rolling basis to one of 4 interventions; After 9/1/2023 design is modified to 3 parallel interventions, with sucralose and aspartame interventions combined into one ASB substitution arm
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to participants' beverage assignment at time of outcome assessment; Investigators will be masked to treatment arm assignments during primary analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Maintain SSBs (Control) (Active Comparator): Instruction to maintain baseline intake of SSBs (months 0-6); then switch to water only (months 6-12)
  Interventions: Behavioral: Maintain usual SSBs; Behavioral: Study app; Behavioral: Beverage delivery
- Substitute Aspartame ASBs (participants randomized through 8/31/2023) (Experimental): Instruction/guidelines to eliminate SSBs and replace, where possible with beverages artificially sweetened with aspartame (months 0-6); then switch to water only (months 6-12)
  Interventions: Behavioral: Substitute to non-SSBs; Behavioral: Study app; Behavioral: Beverage delivery
- Substitute Sucralose ASBs (participants randomized through 8/31/2023) (Experimental): Instruction/guidelines to eliminate SSBs and replace, where possible with beverages artificially sweetened with sucralose (months 0-6); then switch to water only (months 6-12)
  Interventions: Behavioral: Substitute to non-SSBs; Behavioral: Study app; Behavioral: Beverage delivery
- Substitute Water (Experimental): Instruction/guidelines to eliminate SSBs and replace with water (months 0-12)
  Interventions: Behavioral: Substitute to non-SSBs; Behavioral: Study app; Behavioral: Beverage delivery
- Substitute ASBs (participants randomized on or after 9/1/2023) (Experimental): Instruction/guidelines to eliminate SSBs and replace, where possible with beverages artificially sweetened with choice of non-nutritive sweeteners such as sucralose or aspartame
  Interventions: Behavioral: Substitute to non-SSBs; Behavioral: Study app; Behavioral: Beverage delivery

INTERVENTIONS:
Behavioral: Maintain usual SSBs — Instruction/guidelines to maintain baseline intake of SSBs (months 0-6); then switch to water only (months 6-12)
  Arms: Maintain SSBs (Control)
Behavioral: Substitute to non-SSBs — Instruction/guidelines to eliminate SSBs and replace, where possible, with beverages consistent to group assignment (months 0-6); then switch to water only (months 6-12)
  Arms: Substitute ASBs (participants randomized on or after 9/1/2023); Substitute Aspartame ASBs (participants randomized through 8/31/2023); Substitute Sucralose ASBs (participants randomized through 8/31/2023); Substitute Water
Behavioral: Study app — Engage with a motivational mobile app to track beverage intake and complete study data collection
Behavioral: Beverage delivery — Select from approved beverages for a monthly at-home delivery (months 0-6)

SUMMARY:
Sugar-sweetened beverages (SSBs) contribute an alarming ~7% of calories in the US diet among adults, making SSBs the single largest source of added sugar. However, whether artificially sweetened beverages are a healthful alternative for reducing SSB intake among habitual SSB consumers is unknown. Therefore, the investigators will conduct a 4-arm randomized diet intervention trial to test the effects of substituting SSBs with calorie-free alternatives on body weight and health, among habitual SSB consumers with overweight/obesity.

DETAILED DESCRIPTION:
The SUBstituting with Preferred OPtions (SUB-POP) trial, is a parallel-arm randomized controlled trial (RCT) to test the effects of substituting SSBs with non-caloric options on body weight and markers of type 2 diabetes and cardiometabolic health. Eligible adult participants will be randomized to 1 of 4 beverage groups and receive at-home monthly deliveries of beverages for 6 months. In-person clinic visits will be conducted at baseline, 6, and 12 months. After the 6 months of assigned beverage substitution and delivery, all participants will be instructed to substitute SSBs with water only for a final 6-month observational period. In-person clinic visits will collect technician-measured anthropometrics, blood pressure, biospecimen samples (blood, urine, stool [subset]), and assess physical activity, diet, beverage frequency, and taste preference. The SUB-POP app-based assessments and online diet recall will ascertain daily beverage intake, while diet (via 3 24-hour recalls), physical activity, and overall beverage frequency will be collected every 1-3 months. A subset will receive at-home digital scales to transmit daily body weight for energy balance and caloric compensation modeling. SUB-POP is a novel RCT that will enroll adult regular SSB consumers with overweight or obesity to evaluate the effectiveness of substituting SSBs with non-caloric options in a real-world, un-blinded setting. The trial will leverage social media recruitment methods, achieve ≥30% non-White participants, implement innovative intervention delivery, adherence, and data collection tools, and partition the artificially-sweetened beverage (ASB) substitution intervention to the two most common artificial sweetener types (aspartame, sucralose) to explore potential heterogeneity. Whether ASBs, which are largely free of calories and sugar, provide a healthful interim strategy to transition to water among habitual SSB consumers is unknown. Thus, by addressing this large gap in the understanding of how to address a highly prevalent and concerning dietary exposure, the investigators will inform dietary guidelines and clinical recommendations for the prevention of obesity, type 2 diabetes, and cardiometabolic disease risks. The primary outcomes are change in body weight from baseline to 6 months between the 3 beverage substitution groups (aspartame ASBs, sucralose ASBs, and water) vs. the maintain SSBs control group, adjusting for multiple comparisons. The investigators and staff will be blinded to group assignment at outcome assessments. Intention-to-treat analysis will be used.

After 9/1/2023 the 2 ASB intervention groups (sucralose, aspartame) are combined into a single ASB intervention group; participants randomized on or after 9/1/2023 will be randomized to 1 of 3 beverage groups: maintain SSBs (months 0-6; then switch to water months 6-12); switch to ASBs (months 0-6; then switch to water months 6-12); switch to water (months 0-12). The primary outcomes are change in body weight from baseline to 6 months between the 2 beverage substitution groups (ASBs [all ASB intervention groups combined] and water) vs. the maintain SSBs control group, adjusting for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20-69 years
2. Consume ≥1 serving/day (12 oz.) of SSBs (SSBs include soda, fruit drinks, energy drinks, sports drinks, and sweetened waters, sweetened with high fructose corn syrup, sucrose, or fruit juices. SSBs do not include 100% fruit juice, sweetened teas, or flavored milk.)
3. BMI 25.0 to 45.0 kg/m2
4. Access to a smartphone and willingness and ability to download study app
5. Willing to consume beverages consistent with any of the 4 possible group assignments for 6 months

Exclusion Criteria:

1. Physician diagnosis of T2D or fasting glucose ≥126 mg/dL at in-person screening visit
2. Intention to move away from greater Boston area within 1 year from randomization
3. Major medical illness (known cardiovascular disease, cancer, kidney disease, cirrhosis, etc.)
4. Phenylketonuria (PKU)
5. Medication that may affect weight or other study endpoints
6. Another family or household member participating in the study
7. Pregnant in the past 12 months, currently breastfeeding, or planning to become pregnant during the study period

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Weight Change at 6 months | Baseline, Month 6
  Change in total body weight calculated as the month 6 weight minus the baseline weight

SECONDARY OUTCOMES:
Waist Circumference Change | Baseline, Month 6
  Calculated as month 6 minus baseline value
Sussex Sweet Taste Preference Score Change (0 to 100 where higher score indicates greater liking of sweet taste) | Baseline, Month 6
  Calculated as month 6 minus baseline value
Beverage Intake Change (oz/d) | Baseline, Month 6
  Calculated as month 6 minus baseline value
Fasting Plasma Glucose Change | Baseline, Month 6
  Calculated as month 6 minus baseline value
Fasting Blood Insulin Change | Baseline, Month 6
  Calculated as month 6 minus baseline value
HOMA-IR Change | Baseline, Month 6
  Calculated as month 6 minus baseline value
HbA1c Change | Baseline, Month 6
  Calculated as month 6 minus baseline value
TG/HDL Ratio Change | Baseline, Month 6
  Calculated as month 6 minus baseline value
Weight Change Sustainability | Baseline, Month 6
  Calculated as month 6 minus baseline value, month 12 minus month 6 value

OTHER OUTCOMES:
Waist Circumference Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Sussex Sweet Taste Preference Score Change (0 to 100 where higher score indicates greater liking of sweet taste) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Total Beverage Intake Change (oz/d) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
SSB Beverage Intake Change (oz/d) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
ASB Beverage Intake Change (oz/d) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Water Intake Change (oz/d) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
HOMA-IR Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Fasting Blood Insulin Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Fasting Plasma Glucose Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
HbA1c Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Triglycerides Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
TG/HDL Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
HDL-C Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
LDL-C Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Blood Pressure (Systolic and Diastolic) Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
hsCRP Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Interleukin-6 Change | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Alternative Healthy Eating Index 2015 Diet Score Change (Scale 0 to 100 with higher score indicating greater adherence to the dietary pattern) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Self-Reported Added Sugar Change (g/d from 24 hour diet recall) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Self Reported Added Sugar Change (%kcal/d from 24 hour diet recall) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Sweets/Desserts Change (serv/d from 24 hour diet recall) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Total Physical Activity Change (MET-hrs/wk) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value
Energy Compensation (kcal/d) Estimated from Repeated Body Weights (Assessed via At-Home Scale) vs. Repeated Energy Intake (Derived from Repeated Self-Reported 24-Hour Diet Recalls) | Baseline, Month 6, Month 12
  Calculated as month 6 minus baseline value, month 12 minus month 6 value

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Tobias, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No